CLINICAL TRIAL: NCT06318299
Title: Effects of Exogenous Ketone Ester Supplementation on 3-hydroxybutyrate Concentrations in Human Cerebrospinal Fluid
Acronym: KetoBrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 109227
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Ketosis
Keywords: Cerebrospinal Fluid; Brain-Derived Neurotrophic Factor; Point-of-Care Testing; Ketone Bodies; Ketone body adminstration
MeSH Terms: conditions — Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone 1 hour (Active Comparator): Ketone ester drink administered one hour before elective lumbar puncture
  Interventions: Dietary Supplement: Ketone Ester
- Ketone 2 hours (Active Comparator): Ketone ester drink administered two hours before elective lumbar puncture
  Interventions: Dietary Supplement: Ketone Ester
- Placebo 1 hour (Placebo Comparator): Placebo drink administered one hour before elective lumbar puncture
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Ester — Commercially available ketone ester drink (KetoneAid, Virginia, USA)
  Arms: Ketone 1 hour; Ketone 2 hours
Other: Placebo — Taste and appearance matched noncaloric placebo drink
  Arms: Placebo 1 hour

SUMMARY:
It is well established that the brain is capable of consuming ketone bodies, especially during low glucose availability, e.g. fasting. Cerebral metabolism of ketone bodies depends on passage of the blood brain barrier and especially the global blood concentration of ketone bodies.

Ketone bodies can be administered exogenously, and the most commonly used in clinical trials is 3-hydroxybutyrate (3-OHB). 3-OHB is carried by simple diffusion and facilitated diffusion through several monocarboxylic acid transporters (MCTs) across the blood-brain barrier.

To our knowledge, no studies in human adults exist that concurrently measure 3-OHB concentrations in blood and cerebrospinal fluid (CSF) after ingestion or infusion of exogenous ketone supplementation, necessitating further study.

Aims:

* The 3-OHB CSF/blood ratio after oral ingestion of 30 g ketone ester - primary endpoint
* The window of effect: Ketone supplementation 1 h or 2 h before CSF sampling
* If concentration measurements by point-of-care testing are non-inferior to mass spectrometry
* If acute 3-OHB ingestion increases plasma brain-derived neurotrophic factor (BDNF) levels

ELIGIBILITY:
Inclusion Criteria:

* All sexes
* Referred to undergo an elective lumbar puncture procedure in the outpatient clinic at Department of Neurology, Aarhus University Hospital.
* Age 18-80 years
* Written and oral consent

Exclusion Criteria:

* Referred to the clinic suspecting severe neuroinflammation
* Special diet habits, including ketogenic diet, fasting, intermittent fasting etc.
* Daily use of insulin or other medication affecting blood glucose and/or glucose metabolism
* Not able to speak or understand Danish and/or give written and oral consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
3-OHB CSF/blood ratio | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink

SECONDARY OUTCOMES:
CSF 3-OHB concentrations, POCT | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink, Point-of-care testing (POCT)
CSF 3-OHB concentrations, Mass Spectrometry | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink, Mass Spectrometry Detection
CSF glucose concentrations | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink
Blood 3-OHB concentrations | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink, Point-of-care testing (POCT)
Plasma 3-OHB concentrations | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink, Mass Spectrometry Detection
Blood glucose concentrations | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink, Point-of-care testing (POCT)
Plasma BDNF concentrations | 1-2 hours after ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink
Blood 3-OHB concentrations | Before ingestion
  Before oral ingestion of 30 g ketone ester drink or placebo drink, Point-of-care testing (POCT)
Plasma 3-OHB concentrations | Before ingestion
  After oral ingestion of 30 g ketone ester drink or placebo drink, Mass Spectrometry Detection
Blood glucose concentrations | Before ingestion
  Before oral ingestion of 30 g ketone ester drink or placebo drink, Point-of-care testing (POCT)
Plasma BDNF concentrations | Before ingestion
  Before oral ingestion of 30 g ketone ester drink or placebo drink

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark